CLINICAL TRIAL: NCT03352323
Title: Evaluation of the Reduction in Erythema by Oxymetazoline Hydrochloride Topical Cream, 1% in Adults With Moderate to Severe Facial Erythema Associated With Rosacea
Brief Title: An Evaluation of the Reduction in Erythema in Adult Patients With Moderate to Severe Persistent Facial Erythema Associated With Rosacea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Padagis LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRG-NY-17-013
Record Dates: First submitted 2017-11-07; First posted 2017-11-24 (Actual); Results first posted 2021-01-05 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Rosacea; Erythema
MeSH Terms: conditions — Rosacea; Erythema | interventions — Oxymetazoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- oxymetazoline cream (Experimental)
  Interventions: Drug: Oxymetazoline

INTERVENTIONS:
Drug: Oxymetazoline — RLD

SUMMARY:
the study will measure the decrease in redness on the face of rosacea subjects

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating female, 18 years of age or older.
2. Signed informed consent form that meets all criteria of current Food and Drug Administration regulations.
3. Females of childbearing potential must not be pregnant or lactating.
4. Females of childbearing potential must agree to the use of a reliable method of contraception throughout the study.
5. Have clinical diagnosis of rosacea with persistent (non-transient) facial erythema.
6. Have < 3 inflammatory lesions on the face.
7. Have an erythema score of 3 (moderate) or 4 (severe) for both the CEA and the PSA that is reflective of the overall targeted areas.
8. Willing to minimize external factors that might trigger rosacea flare-ups (e.g., spicy foods, hot drinks, hot environments, prolonged sun exposure, strong winds, emotional stress and alcoholic beverages) during the study.

Exclusion Criteria:

1. Forms of rosacea that, in the opinion of the Investigator, would interfere with the diagnosis or assessment of study endpoints
2. Patient has a skin condition that, in the opinion of the Investigator, would interfere with the diagnosis or assessment of rosacea
3. Patients with active sunburn or excessive facial hair such as beards, sideburns, moustaches, etc.
4. Patients with moderate to severe telangiectasial masses
5. History of blood dyscrasia.
6. Significant history or current evidence of any uncontrolled chronic or serious disease or medical condition that would, in the judgment of the Investigator, would put the subject at undue risk or compromise the study assessments.
7. History or current evidence of Raynaud's syndrome, severe, unstable or uncontrolled cardiovascular disease, orthostatic hypotension, uncontrolled hypertension or hypotension, thromboangiitis obliterans, cerebral or coronary insufficiency, renal or hepatic or renal impairment, scleroderma, Sjögren's syndrome, depression, or narrow-angle glaucoma to an extent that, in the opinion of the Investigator, would place the subject at undue risk.
8. Female patients taking hormonal contraceptives or oral estrogen for less than one month or those that plan to change the dosage regimen during the course of the study.
9. Previous participation in this study.
10. Employees of the Investigator or research center or their immediate family members.
11. Inability to understand the requirements of the study and the relative information and are unable or not willing to comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- J&S Studies, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxymetazoline Cream: Rhofade cream
Period: Overall Study
Arm/Group | Oxymetazoline Cream
Started | 50
Completed | 49
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Oxymetazoline Cream
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (15.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 50
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Responder
Description: Responder is defined as a 2-grade improvement from pre-dose on Day 1 on both the Clinician Erythema Assessment and Patient Self Assessment scales
Time Frame: Day 15
Population: Per-protocol population used for analysis; one subject was not compliant with drug applications
Measure: Number; unit: percentage of responders
Arm/Group | Oxymetazoline Cream
Number analyzed (Participants) | 48
percentage of responders | 16.7

ADVERSE EVENTS:
Time Frame: 15 days
Arm/Group | Oxymetazoline Cream
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 3/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxymetazoline Cream (N=50)
Headache (Nervous system disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/23/NCT03352323/Prot_001.pdf
  • Statistical Analysis Plan (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/23/NCT03352323/SAP_000.pdf